CLINICAL TRIAL: NCT04587765
Title: Effect of Extra-curricular Sports Activities After School on Primary School Children's Academic Performance in China: A Non-inferiority Cluster Randomized Controlled Trial
Brief Title: Effect of Extra-curricular Sports Activities After School on Primary School Children's Academic Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SYSU-OPH-008
Record Dates: First submitted 2020-10-02; First posted 2020-10-14 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Extra-curricular Sports
Keywords: academic performance; physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: open,non-inferiority cluster randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extra sports group (Experimental): The group follows the schedule of school teaching programme. Extra-curricular sports classes will be organized and provided in this group of schools in the afternoon after school until 6 p.m. (Monday to Friday).
  Interventions: Behavioral: Extra-curricular sports
- Conventional group (No Intervention): The group follows the schedule of school teaching programme. Students arrange their own after-school time after school.

INTERVENTIONS:
Behavioral: Extra-curricular sports — The group follows the schedule of school teaching programme. Extra-curricular sports classes will be organized and provided in this group of schools in the afternoon after school until 6 p.m. (Monday to Friday).
  Arms: Extra sports group

SUMMARY:
The process of urbanization and the rapid development of information technology have greatly reduced the space and time available for children's outdoor activities. In this study, we expect to study the effects of the addition of physical education classes after school on the academic performance, mental health, physical fitness, and myopia among primary school children.

DETAILED DESCRIPTION:
Urbanization has led to a shrinking of the space suitable for residential activities and a dramatic change in the behavioural patterns, which is particularly evident in children. The spread and development of information technology has reduced children's time for physical activity. Previous studies have found that physical activity is essential for the growth and development of adolescents, preventing and reducing obesity, slowing the development of myopia, and is closely linked to mental health. However, parents in China are concerned that increased outdoor activity will reduce the amount of time spent studying and affect academic performance. Currently, there is a lack of strong evidence on the impact of physical activity on academic performance. In this study, we propose to provide after-school physical education classes for students in primary schools in a rapidly urbanizing area, and assess the effects of the intervention on children's academic performance, physical fitness, myopia, and mental health to provide evidence for the development of educational programs and arrangements for after-school activities.

ELIGIBILITY:
Inclusion Criteria:

1. Pupils in the third and fourth grades of primary schools in Yudu County;
2. Voluntary participation in this study with consent and informed consent signed by guardians.

Exclusion Criteria:

* Exclusion criteria for school

  1. Lack of a third or fourth grade;
  2. Average class size less than 30 students;
  3. No conditions for two classes to play sports at the same time.
* Exclusion criteria for students 4. Two or more days Monday to Friday not available to participate in studies under the project programme; 5. Unsuitability for health or physical reasons to participate in sports activities; 6. Refusal to sign informed consent.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2032 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Mathematics test scores at the end of the first academic year | 1 year
  The test paper will follow the design principles of International Mathematics and science learning, and referring to the local unified examination papers of grade three and grade four, the unified examination questions are formulated to evaluate the students' learning in school

SECONDARY OUTCOMES:
Combined physical fitness test score at the end of the first academic year | 1 year
  Total scores of physical fitness tests according to 2018 National Physical Fitness Survey Monitoring Programme
Incidence of myopia in the first school year | 1 year
  Spherical equivalent after mydriasis ≤ -0.5 D in either eye
Happiness Assessment at the end of the first academic year | 1 year
  Happiness score is rated by Chinese version of the WHO-5 including 5 items with ratings: 0, at no time-5, all of the time. The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being
Mathematics test scores at the end of the second school year | up to 2 years
  The test paper will follow the design principles of International Mathematics and science learning, and referring to the local unified examination papers of grade three and grade four, the unified examination questions are formulated to evaluate the students' learning in school
Combined physical fitness test scores at the end of the second academic year | up to 2 years
  Total scores of physical fitness tests according to 2018 National Physical Fitness Survey Monitoring Programme
Cumulative incidence of myopia over two school years | up to 2 years
  Spherical equivalent after mydriasis ≤ -0.5 D in either eye
Happiness assessment at the second school year | up to 2 years
  Happiness score is rated by Chinese (September, 2007) version of the WHO-5 including 5 items with ratings: 0, at no time-5, all of the time. The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being
Satisfaction assessment | 1 year
  Satisfaction of pupils in the intervention group with the addition of PE after school will be measured by a questionnaire which is designed by reaserchers.

CONTACTS AND LOCATIONS:
Overall Officials: Yangfa Zeng, Master, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Yudu, Ganzhou, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nunes HEG, Silva DAS, Goncalves ECA. Prevalence and factors associated with stages of behavior change for physical activity in adolescents: a systematic review. World J Pediatr. 2017 Jun;13(3):202-209. doi: 10.1007/s12519-017-0027-4. Epub 2017 Mar 22. PMID 28332101
- [Background] Cai Y, Zhu X, Wu X. Overweight, obesity, and screen-time viewing among Chinese school-aged children: National prevalence estimates from the 2016 Physical Activity and Fitness in China-The Youth Study. J Sport Health Sci. 2017 Dec;6(4):404-409. doi: 10.1016/j.jshs.2017.09.002. Epub 2017 Sep 6. PMID 30356639
- [Background] He M, Zeng J, Liu Y, Xu J, Pokharel GP, Ellwein LB. Refractive error and visual impairment in urban children in southern china. Invest Ophthalmol Vis Sci. 2004 Mar;45(3):793-9. doi: 10.1167/iovs.03-1051. PMID 14985292
- [Background] Gray C, Gibbons R, Larouche R, Sandseter EB, Bienenstock A, Brussoni M, Chabot G, Herrington S, Janssen I, Pickett W, Power M, Stanger N, Sampson M, Tremblay MS. What Is the Relationship between Outdoor Time and Physical Activity, Sedentary Behaviour, and Physical Fitness in Children? A Systematic Review. Int J Environ Res Public Health. 2015 Jun 8;12(6):6455-74. doi: 10.3390/ijerph120606455. PMID 26062039
- [Background] Grgic J, Dumuid D, Bengoechea EG, Shrestha N, Bauman A, Olds T, Pedisic Z. Health outcomes associated with reallocations of time between sleep, sedentary behaviour, and physical activity: a systematic scoping review of isotemporal substitution studies. Int J Behav Nutr Phys Act. 2018 Jul 13;15(1):69. doi: 10.1186/s12966-018-0691-3. PMID 30001713
- [Background] French AN, Morgan IG, Mitchell P, Rose KA. Risk factors for incident myopia in Australian schoolchildren: the Sydney adolescent vascular and eye study. Ophthalmology. 2013 Oct;120(10):2100-8. doi: 10.1016/j.ophtha.2013.02.035. Epub 2013 May 11. PMID 23672971
- [Background] He M, Xiang F, Zeng Y, Mai J, Chen Q, Zhang J, Smith W, Rose K, Morgan IG. Effect of Time Spent Outdoors at School on the Development of Myopia Among Children in China: A Randomized Clinical Trial. JAMA. 2015 Sep 15;314(11):1142-8. doi: 10.1001/jama.2015.10803. PMID 26372583
- [Background] Biddle SJ, Asare M. Physical activity and mental health in children and adolescents: a review of reviews. Br J Sports Med. 2011 Sep;45(11):886-95. doi: 10.1136/bjsports-2011-090185. Epub 2011 Aug 1. PMID 21807669
- [Background] Alvarez-Bueno C, Pesce C, Cavero-Redondo I, Sanchez-Lopez M, Garrido-Miguel M, Martinez-Vizcaino V. Academic Achievement and Physical Activity: A Meta-analysis. Pediatrics. 2017 Dec;140(6):e20171498. doi: 10.1542/peds.2017-1498. PMID 29175972
- [Derived] Wang D, Xiong R, Zhang J, Han X, Jin L, Liu W, Qu Y, Chen Q, Chen S, Chen X, Li Y, He M, Zeng Y, Liu Y. Effect of Extracurricular After-School Physical Activities on Academic Performance of Schoolchildren: A Cluster Randomized Clinical Trial. JAMA Pediatr. 2023 Nov 1;177(11):1141-1148. doi: 10.1001/jamapediatrics.2023.3615. PMID 37721735